CLINICAL TRIAL: NCT03425968
Title: Lower Extremity Alignment and Dynamic Control With Associated Injury Risk in College Athletes With Knee Hyperextension
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM106052E
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Knee Hyperextension
Keywords: Injury rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee hyperextension group: athletes who has knee hyperextension
- Control group: athletes who doesn't have knee hyperextension

SUMMARY:
Knee hyperextension, also called genu recurvatum or back knee, is commonly seen in women, people with ligamentous laxity, stroke and cerebral palsy patients. This faulty posture would result in excessive tension of the passive tissues such as anterior cruciate ligament (ACL) and posterior capsule of the knee. Subjects may also develop compensations at hip and ankle joint, as well as lower extremity malalignment. Muscles surrounding the knee could also become dysfunctional when performing functional tasks requiring stability during terminal knee extension, during which uncontrolled knee hyperextension could easily be utilized to lock the joint for stability in gait and stair climbing. In athletes, landing from a jump on an extended knee is one of the common reasons resulting in ACL injury. Little is known about the injury rate of athletes with knee hyperextension who participate in sports involving jump-landing activities.

The aim of the study is to explore if knee hyperextension is associated with poor lower extremity alignment and dynamic control and injury rate in athletes requiring jump-landing activities.

One of the study hypothesis is that athlete with knee hyperextension can find more compensatory lower extremity alignments and poor control in dynamic movement than control group.

The other hypothesis is with or without knee hyperextension, the parameter of lower extremity alignment and dynamic control can predict injury rate in jump landing athlete.

DETAILED DESCRIPTION:
Investigators expect to recruit 100 subjects into 2 group- control group and knee hyperextension group (KH group). In knee hyperextension group, investigators will include college athletes having knee hyperextension alignment, no lower extremity injuries in past three months, and participating in jump-landing activities. Control group will match the gender, age, height, weight and sports to KH group. Inclusion criteria is the same as KH group, except the knee hyperextension angle is <5⁰ in control group. Every subjects will receive the first time assessment and follow up by filling the injury-follow-up form every months for about four months.

At the first assessment, investigators will measure lower extremity alignments include pelvic angle in sagittal plane, hip anteversion, tibiofemoral angle, knee hyperextension angle in supine and standing position, tibial rotation angle, and navicular drop; lower extremity muscle flexibility include rectus femoris, hamstrings, gastrocnemius, soleus, iliotibial band; lower extremity muscle strength include hip, knee, muscle group; dynamic control task will record tibio-femoral acceleration, angle change ground reaction force and EMG muscle firing during vertical jump and drop jump.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20 years old
* knee hyperextension ≥ 5⁰
* participate in jump- landing sports
* training at least 3 days per week
* no lower extremity injury last 3 months

Exclusion Criteria:

* having knee surgery before
* In the past three months have occurred lower extremity musculoskeletal injury leading the person can't participate in training or competition for at least three days

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: college athletes in Yang-Ming University and University of Taipei
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Injury type | 4 months
  Record injury type
Injury duration | 4 months
  time loss during the game or training (days)

SECONDARY OUTCOMES:
Lower extremity alignments-pelvic tilt on sagittal plane | 1st day
  pelvic tilt on sagittal plane in degree
Lower extremity alignments-hip anteversion | 1st day
  hip anteversion in degree
Lower extremity alignments-tibiofemoral angle | 1st day
  tibiofemoral angle in degree
Lower extremity alignments-knee hyperextension angle | 1st day
  knee hyperextension angle in supine and standing posture in degree
Lower extremity alignments-tibial rotation angle | 1st day
  tibial rotation angle in degree
Lower extremity alignments-hip external rotation angle | 1st day
  hip external rotation angle in degree
Lower extremity alignments-hip internal rotation angle | 1st day
  hip internal rotation angle in degree
Lower extremity alignments-navicular drop | 1st day
  navicular drop normalized with foot length in %
Rectus femoris flexibility | 1st day
  measure knee angle in prone knee bend position
Hamstrings flexibility | 1st day
  measure knee angle in 90-90 straight leg raise test
Gastrocnemius flexibility | 1st day
  measure ankle dorsiflexion angle in standing position without rearfoot lift off the floor
Soleus flexibility | 1st day
  measure ankle dorsiflexion angle in knee flex standing position without rearfoot lift off the floor
Iliotibial band flexibility | 1st day
  use Ober's test to measure the angle below horizontal level
Dynamic task parameters-acceleration and angle | 1st day
  anteroposterior acceleration and angle changes at knee joint
Dynamic task parameters-ground reaction force | 1st day
  ground reaction force
Dynamic task parameters-Electromyography (EMG) | 1st day
  use EMG to detect muscle firing during jump task
knee extensors muscle strength | 1st day
  knee extensors by hand held dynamometer
knee flexors muscle strength | 1st day
  knee flexors by hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yin Chen, PhD, Principal Investigator — National Yang-Ming University The Department of Physical Therapy and Assistive Technology
Locations (1):
- National Yng Ming University, Taipei, 北投區, Taiwan